CLINICAL TRIAL: NCT03530852
Title: A 90 Day, Phase 3, Open Labeled Exploratory Study of RELiZORB to Evaluate Safety, Tolerability, and Nutrient Absorption in Children With Short Bowel Syndrome Who Are Dependent on Parenteral Nutrition
Brief Title: A 90 Day, Phase 3,Open Labeled Exploratory Study of RELiZORB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Alcresta Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Puder, MD, PhD, Professor Pediatric General Surgery, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00028297
Record Dates: First submitted 2018-04-13; First posted 2018-05-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Short Bowel Syndrome; Malabsorption
MeSH Terms: conditions — Short Bowel Syndrome; Malabsorption Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Relizorb treatment (Experimental): Patients will have tube feeds placed through chamber and evaluate wean from parenteral nutrition
  Interventions: Device: Relizorb

INTERVENTIONS:
Device: Relizorb — Tube feeds run across device to digest fats.

SUMMARY:
Children with inadequate intestinal absorption due to loss of large amounts of small bowel require intravenous nutrition (feeding through the vein) to sustain hydration and nutrition to avoid starvation and dehydration; however, intravenous (IV) nutrition can lead to complications including liver failure. Tube feeding directly to the small intestine avoids the complications of IV nutrition, but fats are not fully digestible due to inadequate bowel function. We propose to predigest the fat using a small cartridge attached to the feeding tube to allow for rapid absorption with the possibility of reducing or eliminating the need for intravenous nutrition

DETAILED DESCRIPTION:
Project Summary/Abstract

Short bowel syndrome (SBS) is often due to the loss of large amounts of small intestine that compromises digestive absorption. The treatments include (1) a high-calorie diet that includes vitamins, minerals, carbohydrates, proteins and fats; (2) injections of vitamins and minerals; (3) administration of drugs to slow the normal movement of the intestine or to increase the surface area of the intestinal lining; and (4) feeding through the vein (i.e., parenteral nutrition or PN). Many patients cannot wean from PN due to reduced intestinal length or function. Patients on long-term PN frequently experience serious metabolic complications, sepsis, hepatic biliary disorders including cholestasis, and fibrosis and can progress to liver failure. Full intestinal feeding (enteral nutrition) without PN is the optimal way to prevent the above complications.

Enterally administered long chain triglycerides in patients with SBS, especially those with hepatic dysfunction, are not well tolerated due to bile acid malabsorption, which leads to decreased micelle formation and fat digestion. The dietary fat is unable to be emulsified by the bile acids and acted on by lipases before exiting the patient as stool. Switching to other forms of fat such as medium-chain triglycerides (MCTs) that do not require micelles for absorption may be better tolerated in patients with bile acid or pancreatic insufficiency but are not optimal as they increase the osmotic load in the intestine. This may increase the chance of stool dumping; moreover, MCTs do not contain essential fatty acids (FAs). The ability to provide the essential FAs such as those present in enteral formulas in a form that does not require the formation of micelles for absorption, would allow patients with SBS and those who are no longer PN dependent to receive adequate nutrition and continue to maintain the same growth trajectory as when they received the majority of their nutrition parenterally.

RELiZORB is a digestive enzyme cartridge connected in-line with enteral feed tubing sets designed to mimic the function of pancreatic lipase. It is hypothesized that by using an external lipase device (RELiZORB) enteral nutrition will be better absorbed, and PN dependence reduced as enteral autonomy is increased. This product uniquely eliminates the need for intestinal emulsification and lipase activity and eliminates the risk of drugs, including lipases, allowing absorption at the time the diet enters the gut. The device has been shown to digest >90% of fat in most enteral formulas.

This is a phase 3, open label single center clinical trial to determine the safety, tolerability, and bioavailability of the RELiZORB enzyme cartridge with enteral nutrition when used daily for 90 days in pediatric subjects with SBS, aged 2 years - 18 years, who are PN dependent. The change in PN calories from baseline, assessed at Day 7, 14, 28, 60, and 90, will be assessed by area under the curve and presented with a 95% confidence interval. The number (percent) of treatment-emergent adverse events, grade 2 or above, will be tabulated. Changes in growth, fecal fat, plasma FAs, PN volume, and enteral/oral nutrition will be described.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, ages 2 years to 18 years, inclusive.
2. Diagnosed with SBS, as determined by medical history and PN dependence (i.e. need for PN for >60 days after intestinal resection or a bowel length <25% of expected).
3. Congenital or acquired gastrointestinal disease requiring surgical intervention that has occurred at least 3 months prior to screening.
4. Patient is on parenteral lipid and at least 30% of daily caloric and fluid intake has been provided by PN for a least 6 months prior to screening
5. Stable PN nutrition requirement, determined by less than 5% reduction in PN nutrition calories for at least 1 month prior to screening, or at the discretion of the investigator.
6. Screening direct bilirubin that is in the normal range for age and is not determined to be clinically significant by the investigator.
7. Subject has an existing feeding tube, is receiving enteral nutrition via a pump at a rate>10ml/hr but <120ml/hr, and is able to tolerate at least 10 ml/kg/day enteral nutrition.
8. Stable enteral nutrition requirement with no change in formula composition or rate for at least 1 month prior to screening.
9. The parent or legal guardian of the patient is able to read, understand, and is willing to provide informed consent (and assent, if applicable).
10. The patient (if assent is applicable) or parent or legal guardian of the patient is able to understand the requirements of the study and is willing to bring the patient to all clinic visits and complete all study related procedures (as determined by the investigator).

A parent or legal guardian is willing to provide written authorization for the use and disclosure of protected health information.

Exclusion criteria:

1. Other causes of chronic liver disease other than SBS (i.e., hepatitis C, cystic fibrosis, biliary atresia, alpha 1 anti-trypsin deficiency, and Alagille syndrome).
2. The patient has had a bowel lengthening procedure, including but not limited to, a STEP procedure.
3. Any serum triglyceride concentration >400 mg/dL at screening.
4. Pancreatic insufficiency as defined as the use of pancreatic enzymes within 30 days prior to screening.
5. Evidence of untreated intestinal obstruction or active stenosis, as determined by the investigator.
6. Unstable absorption due to cystic fibrosis or known DNA abnormalities (i.e., familial adenomatous polyposis, Fanconi syndrome) as determined by the investigator.
7. History of microvillus inclusion disease, as determined by medical history.
8. Severe known dysmotility syndrome (i.e., pseudo-obstruction, gastroschisis-related motility disorders), as determined by the investigator.
9. Initiation of teduglutide or other GLP-2 analogues within 6 months of screening
10. Use of growth hormone, or supplemental glutamine within 3 months prior to screening.
11. Use of cisapride within 30 days prior to screening.
12. Active clinically significant pancreatic or biliary disease, as determined by the investigator.
13. Patients are receiving formulas that are not compatible with the RELiZORB cartridge (example, insoluble fiber-containing formulas)
14. Determined by the investigator to be unsuitable for participation for any reason.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the RELiZORB enzyme cartridge on the absorption of enteral nutrition based on PN calories | 90 days
  To determine the effectiveness of the RELiZORB enzyme cartridge on the absorption of enteral nutrition when used daily for a total 90 days of treatment, in pediatric subjects with SBS who are PN dependent, aged 2 years - 18 years, by measuring the change in PN calories from baseline, assessed at days 7, 14, 28, 60, and day 90. Each subject will be on the study for a total of 90 days.

SECONDARY OUTCOMES:
Effectiveness of the RELiZORB enzyme cartridge on the absorption of enteral nutrition based on body weight change | 90 days
  To determine the effectiveness of the RELiZORB enzyme cartridge on the absorption of enteral nutrition when used daily for a total 90 days of treatment, in pediatric subjects with SBS who are PN dependent, aged 2 years - 18 years, by measuring the change in body weight from baseline, assessed at days 7, 14, 28, 60, and day 90. Each subject will be on the study for a total of 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Puder, MD, PhD., Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Freedman S, Orenstein D, Black P, Brown P, McCoy K, Stevens J, Grujic D, Clayton R. Increased Fat Absorption From Enteral Formula Through an In-line Digestive Cartridge in Patients With Cystic Fibrosis. J Pediatr Gastroenterol Nutr. 2017 Jul;65(1):97-101. doi: 10.1097/MPG.0000000000001617. PMID 28471913
- [Derived] Tsikis ST, Fligor SC, Mitchell PD, Hirsch TI, Carbeau S, First E, Loring G, Rudie C, Freedman SD, Martin CR, Gura KM, Puder M. Fat digestion using RELiZORB in children with short bowel syndrome who are dependent on parenteral nutrition: Protocol for a 90-day, phase 3, open labeled study. PLoS One. 2023 Mar 1;18(3):e0282248. doi: 10.1371/journal.pone.0282248. eCollection 2023. PMID 36857339